CLINICAL TRIAL: NCT03385733
Title: The Effects of Inspiratory Muscle Training on Exercise Capacity, Physical Activity and Quality of Life in Pulmonary Hypertension
Brief Title: Inspiratory Muscle Training in Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Biruni University (Other)
Responsible Party: Principal Investigator, Goksen Kuran Aslan, Associated Proff., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAslan; BuketA (Other: BiruniU)
Record Dates: First submitted 2017-12-21; First posted 2017-12-28 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; inspiratory muscle training; functional capacity; physical activity
MeSH Terms: conditions — Hypertension, Pulmonary; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients will randomize into two groups as Group A: inspiratory muscle training, and Group B (control group)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training group (Experimental): Patients will continue 8 weeks, 5 days, 2 times 15 minutes training program with %30 MIP at home.
  Interventions: Other: inspiratory muscle training
- control group (No Intervention): Patients will continue 8 weeks, 5 days, 2 times 15 minutes training program with 9 cmH2O pressure at home.

INTERVENTIONS:
Other: inspiratory muscle training — The treatment group received IMT. Patients were trained using an inspiratory threshold-loading device
  Arms: Inspiratory muscle training group

SUMMARY:
The aim of this study is to investigate the effective of inspiratory muscle training on respiratory function, exercise capacity, physical activity and quality of life.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a condition which is seen with hemodynamic differences, pulmonary vascular resistance and right heart failure. Patients with pulmonary hypertension have, dyspnea, physical inactivity, reduced condition and respiratory muscle dysfunction. Aerobic exercise programs in patients with pulmonary hypertension are reported to result in improved exercise capacity and endurance of the patients, improvement in WHO functional class and quality of life, increased peak workload and increased peripheral muscle function. In recent years, few studies have investigated the efficacy of inspiratory muscle training in patients with PH.The aim of this study is to investigate the effective of inspiratory muscle training on respiratory function, exercise capacity, physical activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Pulmonary Hypertension,
* NYHA functional class I-IV
* MIP pressure <80 cm h2O

Exclusion Criteria:

* COPD
* Conditions which can limit the assessments
* Insufficient cooperation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
mouth pressures | 10 minutes
  MIP and MEP

SECONDARY OUTCOMES:
International Physical Activity Questionnaire-Short Form | 10 minutes
  Physical activity
Minnesota Living with Heart Failure Questionnaire | 15 minutes
  quality of life
Activity monitoring (Sense wear® Armband) | 3 days
  Metabolic holter
6 minute walking test | 15 minutes
  functional capacity

CONTACTS AND LOCATIONS:
Overall Officials: Goksen Kuran Aslan, Study Director — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Results of the study will share with other researchers